CLINICAL TRIAL: NCT00000229
Title: Buprenorphine Detox With Two Types of Treatment. BBD II
Brief Title: Buprenorphine Detox With Two Types of Treatment. BBD II - 11
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-06969-11; R01DA006969 (NIH); R01-06969-11
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 1996-09

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to compare overall treatment outcome between behavioral versus enhanced behavioral treatment types.

ELIGIBILITY:
Please contact site for information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1995-10

PRIMARY OUTCOMES:
Drug use
Retention
Weeks abstinent
Weeks continuous abstinence
Overall treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States